CLINICAL TRIAL: NCT01741779
Title: The Effect of Diet and Whole-body Vibration Training on Cardiovascular and Autonomic Function in Obese Postmenopausal Women
Brief Title: Diet and Whole-body Vibration Training on Cardiovascular and Autonomic Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Nutrisystem, Inc. (Industry)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSC2011.6728
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Obesity; Pre-hypertension; Hypertension
Keywords: whole body vibration training; hypocaloric diet; prehypertension; hypertension; obesity; arterial function; arterial stiffness; pulse wave velocity; autonomic function; endothelial function; adipocytokines
MeSH Terms: conditions — Obesity; Prehypertension; Hypertension | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hypocaloric diet (Experimental): This arm involves 12 wk of the standard Nutrisystem foods plan complemented by fresh produce and dairy. Subjects consume breakfast, lunch, dinner, and one (women) or two (men) snacks per day.
  Interventions: Other: Hypocaloric diet
- Control (No Intervention): This arm involves not making any change to the subject's lifestyle at the moment of the start of the intervention and for 12 wk.
- Whole body vibration training & diet (Experimental): Lower-body exercise training on a vibration platform and diet
  Interventions: Other: Whole body vibration training & diet
- Whole body vibration training (Experimental): Lower-body exercises 3 times per wk for 12 wk in a vibration platform
  Interventions: Other: Whole Body Vibration Training

INTERVENTIONS:
Other: Whole Body Vibration Training — The Whole body vibration training intervention consists of lower-body exercise in a vibration platform 3 times per wk for 12 wk. The subjects will perform static and dynamic exercises for the legs on the vibration platform. Dynamic exercises will be performed with slow controlled movements starting from an upright position into a 60 degree knee flexion (squat) and maximal heel elevation (toestand). Static exercises will be performed without movement in the joint angles described previously. The training volume will increase progressively over the 12-week training period by increasing the intensity of vibration, duration of the exercise set (30-60 sec), number of sets per exercise, and total duration of the training session, and decreasing the duration of rest periods (30-60 sec).The intensity of vibration and amplitude will also be increased progressively (25-30 Hz of frequency and from low to high amplitude).
  Arms: Whole body vibration training
Other: Hypocaloric diet — The hypocaloric diet intervention consists of 12 wk of the standard Nutrisystem foods plan complemented by fresh produce and dairy. Subjects consume breakfast, lunch, dinner, and one (women) or two (men) snacks per day.
  Arms: Hypocaloric diet
Other: Whole body vibration training & diet — Combination of whole body vibration training and hypocaloric diet
  Arms: Whole body vibration training & diet

SUMMARY:
Obesity is a major risk factor for premature arterial abnormalities including high blood pressure and increased stiffness. Previous studies have shown that weight loss via lifestyle modifications is associated with a decrease in large artery (aorta) stiffness. However, along with decreases in fat mass, hypocaloric diet reduces muscle mass. Whole body vibration results in similar increases in muscle mass and strength than those observed after resistance exercise and is feasible for special populations such as the obese and the elderly.

The investigators hypothesis is that weight loss via diet combined with whole body vibration training would additively reduce arterial stiffness and blood pressure in obese women. The investigators also hypothesize that the improved arterial function with weight loss would be associated with beneficial changes in the main mechanisms involved in BP regulation.

DETAILED DESCRIPTION:
The purpose of the study is to examine the effects of 12 weeks of whole body vibration training (WBVT) and diet on arterial function, autonomic function, and body composition in obese women. Specific aims of the study are to:

To evaluate the extent to which diet and (WBVT) will improve body composition assessed by changes in fat mass and lean mass using dual-energy x-ray absorptiometry and waist circumference.

To investigate that combined diet and (WBVT) are more efficacious than either treatment alone in ameliorating cardiovascular disease risk factors by assessing arterial stiffness (aortic, systemic, and leg), aortic BP and wave reflection, and autonomic function (heart rate variability, vascular sympathetic activity [low-frequency power of systolic BP variability], and baroreflex sensitivity). Flow mediated dilation and circulating levels of adipocytokines (adiponectin and leptin) and endothelial-derived vasodilators (NO metabolites [NOx], 6-keto PGFIa, insulin, and ghrelin) and vasoconstrictors (endothelin-1 [ET-1],8-iso PGF2a,vascular endothelium growth factor [VGEF]) will be assessed as secondary outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 45 to 65 years of age
* At least 1 year after menopause
* Body mass index of 27-39.9
* Sedentary or low active (less than 2 hr per wk)

Exclusion Criteria:

* Younger than 45 or older than 65 years of age
* Body mass index lower than 27, or 40 or higher
* Physically active or competitively active
* Smoker
* Use of hormone replacement therapy of less than 1 yr
* Use of calcium channel blocker or beta blockers
* Use dietary supplementations (e.g.,L-arginine,L-citrulline,antioxidants)
* Uncontrolled diabetes
* Any restriction that would significantly interfere with compliance with the diet (e.g., allergy to nuts or dairy, or need to avoid soy)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Body Composition | 12 weeks
  By measuring fat mass and lean soft tissue mass from dual-energy x-ray absorptiometry and waist circumference
Blood pressure | 12 weeks
  Non-invasive measures of brachial and aortic blood pressure
Arterial Stiffness | 12 weeks
  Using pulse wave velocity of the aorta, systemic, and legs
Pressure Wave Reflection | 12 weeks
  Using the augmentation index from radial tonometry
Autonomic Function | 12 weeks
  Heart rate variability, vascular sympathetic activity [low-frequency power of systolic BP variability], and spontaneous baroreflex sensitivity will be assessed from electrocardiogram and beat-by-beat digital blood pressure

SECONDARY OUTCOMES:
Endothelial Function | 12 weeks
  By measuring circulating levels of adipocytokines (adiponectin and leptin) and endothelial-derived vasodilators (NOx, 6-keto PGFIa, insulin, and ghrelin)and vasoconstrictors (ET-1 and 8-iso PGF2a, VEGF)

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, M.D., Ph.D, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States